CLINICAL TRIAL: NCT00527033
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled Study in Patients With Symptomatic Overactive Bladder
Brief Title: A Study of YM178 in Patients With Symptomatic Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 178-CL-045
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder, Overactive
Keywords: YM178; Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Oral
  Interventions: Drug: YM178
- 2 (Experimental): Oral
  Interventions: Drug: YM178
- 3 (Experimental): Oral
  Interventions: Drug: YM178
- 4 (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YM178 — Oral
  Arms: 1; 2; 3
Drug: Placebo — Oral
  Arms: 4

SUMMARY:
Examine which dose of YM178 is the best in terms of efficacy, safety and tolerability compared to placebo

DETAILED DESCRIPTION:
To investigate the dose-response relationship of YM178 in terms of efficacy, safety and tolerability, and also the superiority of YM178 over placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 20 years suffering from overactive bladder

Exclusion Criteria:

* Pregnant and breastfeeding women
* Any clinically significant abnormal conditions which in the opinion of the investigator makes the patient unsuitable for the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 842 (Actual)
Dates: Start 2007-09-11 (Actual); Primary Completion 2008-04-03 (Actual); Study Completion 2008-04-03 (Actual)

PRIMARY OUTCOMES:
Overactive bladder symptoms | 12 weeks

SECONDARY OUTCOMES:
Overactive bladder symptoms (QOL) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (5):
- Japan (5):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kanto
  - Kyusyu

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Yamaguchi O, Marui E, Igawa Y, Takeda M, Nishizawa O, Ikeda Y, Ohkawa S. Efficacy and Safety of the Selective beta3 -Adrenoceptor Agonist Mirabegron in Japanese Patients with Overactive Bladder: A Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study. Low Urin Tract Symptoms. 2015 May;7(2):84-92. doi: 10.1111/luts.12053. Epub 2014 Mar 11. PMID 26663687
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=166